CLINICAL TRIAL: NCT02259400
Title: Noninvasive Ventilation Strategies for Early Treatment of RDS in Preterm Infants: An RCT
Brief Title: NIV Strategies for RDS in Preterm Infants. NIV (Non Invasive Ventilation), RDS (Respiratory Distress Syndrome)
Acronym: NIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Collaborators: Vittore Buzzi Children's Hospital (Other); Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Vincenzo Salvo, MD, MD, Neonatal Intensive Care Unit, Pediatric Department, Azienda Ospedaliera Universitaria Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIV/RDS-01
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-01

CONDITIONS: RDS of Prematurity
Keywords: NIV; NSIPPV; BiPAP
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants

ARMS (2):
- NSIPPV group (Active Comparator): The NSIPPV is a conventional modality of mechanical ventilation delivered by the nasal ventilator device Giulia (Ginevri, Rome, Italy), that in noninvasive modality detects the inspiratory effort by means of a pneumotachograph, equipped with a fixed orifice (2 mm in diameter for LBW infants), positioned proximally to the nasal interface. Short bi-nasal prongs (NIV set, Ginevri, Rome, Italy), with different size according to infants'weight, will be used as interface.
  Interventions: Device: NSIPPV
- BiPAP group (Active Comparator): The BiPAP is a modality of noninvasive respiratory support that provides two alternate different levels of CPAP in which the babies can breath spontaneously. The BiPAP will be delivered by the Infant Flow-driver device (Infant Flow System, Vyasis Corp,Yorba Linda, California (CA),USA) and bi-nasal prongs as interface (Vyasis Corp,Yorba Linda, CA,USA) with different size according to infants' weight.
  Interventions: Device: BiPAP

INTERVENTIONS:
Device: NSIPPV — In N-SIPPV, the physician will set : an initial PEEP of 4-6 cmH20; a peak inspiratory pressure (PIP) of 15-20 cmH2O ; an inspiratory time (IT) of 0.3-0.4 seconds; a flow rate of 6-10 L/min and a respiratory rate (RR) of 40 bpm with the lowest FiO2 to maintain a oxygen saturation (SpO2) of 88-93%. Weaning from N-SIPPV will be performed with a reduction of the RR to 15 bpm with a PIP of 10-15 cmH2O and PEEP of 4 cmH2O and will be stopped when the baby will not show signs of RDS and with a fraction of inspired oxygen (FiO2)< 0.3.
  Arms: NSIPPV group
Device: BiPAP — In BiPAP, the physician will set : an initial low CPAP-level of 4-6 cmH20 and high CPAP-level of 8-9 cmH20; a time high of 1 second and a pressure exchange rate of 20 bpm, with the lowest FiO2 to maintain a SpO2 of 88-93%. Weaning will start with a progressive reduction of the set pressure exchange rate ( minimum 15 pressures exchange/min), followed by the reduction of the higher level-CPAP down to 6 cmH20 and lower level-CPAP down to 4 cmH20. BiPAP will be stopped when the baby will not show signs of RDS and with a FiO2 < 0.3.
  Arms: BiPAP group

SUMMARY:
The purpose of this study is to determine whether two different strategies of Non Invasive Ventilation (NIV) have different effect on length and failure of NIV support in preterm infants with respiratory distress syndrome (RDS).

DETAILED DESCRIPTION:
A Randomized Control Trial (RCT) conducted in two tertiary level Neonatal Intensive Care Unit (NICU). Ethical approval is needed. Informed and written consent will be obtained prior the delivery from the parents of the babies before the inclusion in the study. All inborn Very Low Birth Weight (VLBW) infants (Birthweight less than 1500 g and Gestational Age < 32 weeks) with signs of RDS, spontaneously breathing and only supported by nasal-Continuous Positive Airway Pressure (NCPAP) in NICU, will be randomized within the first 2 hours of life to receive two different Non Invasive Ventilation (NIV) strategies: Nasal Synchronized Intermittent Positive Pressure Ventilation (N-SIPPV) or Bilevel Continuous Positive Airway Pressure (BiPAP).

ELIGIBILITY:
Inclusion Criteria:

* All inborn VLBW infants (birthweight less than 1500 g and Gestational Age < 32 wks) with signs of RDS, spontaneously breathing and only supported by N-CPAP, will be randomized within the first 2 hours of life to receive two different Non Invasive Ventilation (NIV) strategies.

Exclusion Criteria:

* Apneic or severely depressed newborns requiring invasive ventilation, within two hours from birth
* Newborns with genetic disease and/or with major congenital malformations
* Newborns for whom it was not obtained informed consent within two hours from birth

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo V Salvo, MD, Principal Investigator — Azienda Ospedaliera Universitaria Policlinico "G Martino" Messina

REFERENCES:
- [Background] Committee on Fetus and Newborn; American Academy of Pediatrics. Respiratory support in preterm infants at birth. Pediatrics. 2014 Jan;133(1):171-4. doi: 10.1542/peds.2013-3442. Epub 2013 Dec 30. PMID 24379228
- [Background] Stevens TP, Harrington EW, Blennow M, Soll RF. Early surfactant administration with brief ventilation vs. selective surfactant and continued mechanical ventilation for preterm infants with or at risk for respiratory distress syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003063. doi: 10.1002/14651858.CD003063.pub3. PMID 17943779
- [Background] Bhandari V. Nasal intermittent positive pressure ventilation in the newborn: review of literature and evidence-based guidelines. J Perinatol. 2010 Aug;30(8):505-12. doi: 10.1038/jp.2009.165. Epub 2009 Oct 22. PMID 19847188
- [Background] Kirpalani H, Millar D, Lemyre B, Yoder BA, Chiu A, Roberts RS; NIPPV Study Group. A trial comparing noninvasive ventilation strategies in preterm infants. N Engl J Med. 2013 Aug 15;369(7):611-20. doi: 10.1056/NEJMoa1214533. PMID 23944299
- [Background] Meneses J, Bhandari V, Alves JG, Herrmann D. Noninvasive ventilation for respiratory distress syndrome: a randomized controlled trial. Pediatrics. 2011 Feb;127(2):300-7. doi: 10.1542/peds.2010-0922. Epub 2011 Jan 24. PMID 21262883
- [Background] Roberts CT, Davis PG, Owen LS. Neonatal non-invasive respiratory support: synchronised NIPPV, non-synchronised NIPPV or bi-level CPAP: what is the evidence in 2013? Neonatology. 2013;104(3):203-9. doi: 10.1159/000353448. Epub 2013 Aug 28. PMID 23989138
- [Background] Ricotti A, Salvo V, Zimmermann LJ, Gavilanes AW, Barberi I, Lista G, Colivicchi M, Temporini F, Gazzolo D. N-SIPPV versus bi-level N-CPAP for early treatment of respiratory distress syndrome in preterm infants. J Matern Fetal Neonatal Med. 2013 Sep;26(13):1346-51. doi: 10.3109/14767058.2013.784255. Epub 2013 Apr 17. PMID 23488612
- [Derived] Salvo V, Lista G, Lupo E, Ricotti A, Zimmermann LJ, Gavilanes AW, Barberi I, Colivicchi M, Temporini F, Gazzolo D. Noninvasive ventilation strategies for early treatment of RDS in preterm infants: an RCT. Pediatrics. 2015 Mar;135(3):444-51. doi: 10.1542/peds.2014-0895. Epub 2015 Feb 9. PMID 25667244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 280 VLBW infants with RDS, delivered before 32 weeks of gestational age and with a birth weight <1500 gr, admitted in two NICUs (C. Arrigo, Children's Hospital, Alessandria, Italy and V. Buzzi, Children's Hospital, Milan, Italy) from January 2010 to December 2012.
Pre-assignment Details: 156 Newborns were excluded from the study: 19 had exclusion criteria, 40 not requiring ventilation support, 35 requiring invasive ventilation, 62 not randomized within 2 hours from birth. 124 newborns needed NIV within 2-h from birth, were randomly allocated to receive either NSIPPV (n=62) or BiPAP (n=62).
Groups:
- NSIPPV Group: The NSIPPV is a conventional modality of mechanical ventilation delivered by the nasal ventilator device Giulia (Ginevri, Rome, Italy), that in noninvasive modality detects the inspiratory effort by means of a pneumotachograph, equipped with a fixed orifice (2 mm in diameter), positioned proximally to the nasal interface. Short bi-nasal prongs (NIV set, Ginevri, Rome, Italy), with different size according to infants'weight, will be used as interface.
  NSIPPV: In N-SIPPV, the physician will set : an initial PEEP of 4-6 cmH20; a peak inspiratory pressure (PIP) of 15-20 cmH2O ; an inspiratory time (IT) of 0.3-0.4 seconds; a flow rate of 6-10 L/min and a respiratory rate (RR) of 40 bpm with the lowest FiO2 to maintain a oxygen saturation (SpO2) of 88-93%. Weaning from N-SIPPV will be performed with a reduction of the RR to 15 bpm with a PIP of 10-15 cmH2O and PEEP of 4 cmH2O and will be stopped when the baby will not show signs of RDS and with a fraction of inspired oxygen (FiO2)< 0.3.
Period: Overall Study
Arm/Group | NSIPPV Group | BiPAP Group
Started | 62 | 62
Completed | 62 | 60
Not Completed | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NSIPPV Group | BiPAP Group | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: WEEKS] — GESTATIONAL AGE
  WEEKS | 28.6 (2.1) | 28.8 (2.2) | 28.7 (2.3)
Age, Customized [Number; unit: participants] — GESTATIONAL AGE SUBGROUPS
  participants
    ≤ 26 wGA | 9 | 9 | 18
    > 26 and ≤29 wGA | 33 | 32 | 65
    > 29 wGA | 20 | 21 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 27 | 25 | 52
SMALL FOR GESTATIONAL AGE [Number; unit: participants] — newborn with a birth weight below the 10th percentile for gestational age
  participants | 14 | 12 | 26
BIRTH-WEIGHT [Mean (Standard Deviation); unit: GRAMS] | 1106 (276) | 1165 (275) | 1135 (289)

OUTCOME MEASURES:

1. Primary Outcome: Duration of NIV Support
Description: DURATION OF NON INVASIVE VENTILATION SUPPORT FOR RDS TREATMENT
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: HOURS
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
HOURS | 89 [61 to 143] | 87 [48 to 134]
Statistical Analysis 1: Comparison: NSIPPV Group vs BiPAP Group; Test type: Non-Inferiority or Equivalence — For the calculation of sample size we used the duration of ventilation as the main primary outcome. As no basic data are available for this population, we were able to retrieve from the database of our two NICUs the duration of ventilation on NIV. We assumed a difference of 24-h between the two groups in the duration of NIV as clinically relevant. We used a confidence level α=0.05; the power level desired was 0.80 and consequently we needed 62 patients for each group; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Failure of NIV Support
Description: NUMBER OF NEWBORNS WHO FAILED WITH NON INVASIVE VENTILATION SUPPORT AND NEEDED INTUBATION AND INVASIVE MECHANICAL VENTILATION.
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 62
participants | 10 | 8

3. Secondary Outcome: Death
Time Frame: 2 month
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 62
participants | 0 | 2

4. Secondary Outcome: Bronchopulmonary Dysplasia (BPD)
Time Frame: 36 weeks of postconceptional age or time of discharge
Population: 2 newborns died in bipap group
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 7 | 7

5. Secondary Outcome: Pneumothorax (PNX)
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 2 | 4

6. Secondary Outcome: Intraventricular Hemorrhage (IVH)
Time Frame: 1 month of life
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 2 | 2

7. Secondary Outcome: Periventricular Leukomalacia (PVL)
Time Frame: 3 month of life
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 2 | 4

8. Secondary Outcome: Retinopathy of Prematurity (ROP)
Time Frame: 3 month of life
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 2 | 3

9. Secondary Outcome: Patent Ductus Arteriosus Requiring Pharmacological Treatment (PDA)
Time Frame: first week of life
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 18 | 14

10. Secondary Outcome: Necrotizing Enterocolitis (NEC)
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 0 | 2

11. Secondary Outcome: Newborns Who Received Multiple Surfactant Doses
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 21 | 18

12. Secondary Outcome: Early Onset Sepsis
Time Frame: 5days from birth
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 13 | 15

13. Secondary Outcome: Late Onset Sepsis
Time Frame: after fifth days of life up 2 month of life
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 60
participants | 21 | 14

14. Secondary Outcome: Death
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | NSIPPV Group | BiPAP Group
Number analyzed (Participants) | 62 | 62
participants | 0 | 2

ADVERSE EVENTS:
Time Frame: During hospitalization
Arm/Group | NSIPPV Group | BiPAP Group
Serious Adverse Events (participants affected / at risk) | 2/62 | 6/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSIPPV Group (N=62) | BiPAP Group (N=62)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4
death (General disorders) | 0 | 2 — death from any cause, also not directly related to ventilation modality failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No